CLINICAL TRIAL: NCT03405337
Title: Evaluation of Patient and Physician Reported Reasons for Switching FVIII Replacement Therapies
Brief Title: Evaluation of Patient and Physician Reported Reasons for Switching Factor VIII Replacement Therapies
Acronym: PARkER
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19529
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- FVIII products (prospective): Qualitative patient/caregiver study:
  Hemophilia A patients/caregivers (N=30) having initiated a FVIII products with improved half-life
  Interventions: Drug: FVIII products; Drug: Conventional FVIII replacement therapies
- Conventional FVIII replacement therapies: Qualitative patient/caregiver study:
  Hemophilia A patients/caregivers (N=30) receiving "conventional" FVIII replacement therapy for at least 6 months who are considering switching to a FVIII product with improved half-life within the next 1 year
  Interventions: Drug: Conventional FVIII replacement therapies
- FVIII products (retrospective): Quantitative physician interview/ chart review study:
  Hemophilia A patients (N=100) who have switched from "conventional" FVIII replacement therapy to FVIII products with improved half-life.
  Interventions: Drug: FVIII products; Drug: Conventional FVIII replacement therapies

INTERVENTIONS:
Drug: FVIII products — Adynovate, Eloctate, Afstyla, Kovaltry
  Groups: FVIII products (prospective); FVIII products (retrospective)
Drug: Conventional FVIII replacement therapies — Advate, Kogenate FS, Helixate, Novoeight, Nuwiq, Recombinate, Xyntha

SUMMARY:
This US study will assess hemophilia A patient characteristics, health history and reasons for switching or not switching from both patient/caregiver and physician perspectives. For this purpose, this research study will include hemophilia A: 1) patients who have switched from conventional therapy to new FVIII products with an improved PK profile. 2) patients who remain on conventional therapy (who have never switched) but have considered switching, including those patients who switched from conventional therapy to new FVIII products with improved pharmacokinetics and then subsequently "switched back" to conventional replacement therapy. In doing so, real world evidence will be obtained from both patient and physician perspectives offering key insights for effective therapeutic management of patients with hemophilia A and to more fully understand what drives patient switching from a patient perspective and a physician perspective.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients/caregivers in the Patient/Caregiver Study:

* Patients with hemophilia A (≥ 18 years of age) or caregivers of children with hemophilia A (≥12-<18 years of age)
* Group 1: Hemophilia A patients/caregivers who have switched to FVIII products with improved half-life for the treatment of hemophilia A during the eligibility period. These patients can also include those who have switched back from FVIII products with improved half-life to conventional FVIII replacement therapy within the Data Collection Period
* Group 2: Hemophilia A patients/caregivers who are considering switching to FVIII products with improved half-life within 12 months of the Start of the Documentation period and have been prescribed prophylaxis regimen of at least 2x/week
* Able to understand, read, write and speak English
* Provide electronic informed consent
* Able to access the Internet for at least 20 minutes per day during the Data Collection Period

Inclusion criteria for physicians:

* At least 60% of time spent in direct patient care
* Board-certified or eligible with a Specialty in Hematology or Hematology-Oncology
* Physicians with a specialty in Hematology-Oncology must have at least 10% of their practice dedicated to treatment of hemophilia
* A minimum of 2 years' experience treating hemophilia A patients

Inclusion criteria for patients in the physician chart study:

* Hemophilia A patients age 12 year and over
* Prior treatment with one of the following FVIII replacement products: Adynovate, Afstyla, Eloctate, or Kovaltry
* Patients that have 12 months of medical chart data available; 6 months on conventional therapy and 6 months after switching to FVIII products with improved half-life.

Exclusion Criteria:

Exclusion criteria for patients/caregivers in the Patient/Caregiver Study:

- Hemophilia A patient initiated FVIII products with improved half-life for the treatment at time of diagnosis with hemophilia A.

Exclusion criteria for physicians:

- Unwilling to comply with the study protocol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Population for the Patient/Caregiver Study:
  Hemophilia A patients/caregivers will be recruited via opt-in patient panels and/or research databases.
  Patients with hemophilia A (≥ 18 years of age) or caregivers of children with hemophilia A (≥12-<18 years of age)
  Study Population for the Physician Chart Study:
  The study population for the physician chart review study will be patients, who initiated FVIII products with improved half-life for the treatment of hemophilia A during the eligibility period. In order to obtain a broad patient population that is representative of real world prescribing; all eligible patients will be included in the study irrespective of the FVIII product with improved half-life received.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
The reasons of patients/caregivers "switch" from conventional FVIII replacement therapy to FVIII products with improved half-life | Up to 6 days
  These patients/caregivers will participate in an asynchronous online discussion forum consisting of predetermined open ended and close ended questions for a series of 6 consecutive days completing approximately 20 minutes' worth of questions per day.
The obstacles of switching among hemophilia A patients who did not switch from conventional therapy to FVIII products with improved half-life but who are open to switching | Up to 6 days
  These patients/caregivers will participate in an asynchronous online discussion forum consisting of predetermined open ended and close ended questions for a series of 6 consecutive days completing approximately 20 minutes' worth of questions per day.
The clinical characteristics of patients who switch from conventional FVIII replacement therapy to FVIII products with improved half-life | Up to 4.5 months
  A retrospective patient medical chart review
The changes of treatment characteristics from 6 months prior to switching compared to 6 months after switching from conventional FVIII replacement therapy to FVIII products with improved half-life | Up to 4.5 months
  A retrospective patient medical chart review
The changes of bleeding related outcomes from 6 months prior to switching compared to 6 months after switching from conventional FVIII replacement therapy to FVIII products with improved half-life | Up to 4.5 months
  A retrospective patient medical chart review
The reasons for switching from conventional FVIII replacement therapy to FVIII products with improved half-life, from the physician perspective | Up to 4.5 months
  A retrospective patient medical chart review

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Whippany, New Jersey, United States